CLINICAL TRIAL: NCT03779737
Title: Muscular Strength and Aerobic Capacity, a Symbiotic Relationship With Birth Weight and Metabolic Risk of Colombian Scholchildren: Study SIMAC
Brief Title: Resistance and Aerobic Training, Relationship With Birth Weight in Colombian Children
Acronym: SIMAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación Oftalmológica de Santander Clínica Carlos Ardila Lulle (Other)
Collaborators: Universidad de Santander (Other); Instituto Colombiano para el Desarrollo de la Ciencia y la Tecnología (COLCIENCIAS) (Other Government)
Responsible Party: Principal Investigator, Paul Anthony Camacho Lopez, Principal Investigator, Fundación Oftalmológica de Santander Clínica Carlos Ardila Lulle
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 651765741093
Record Dates: First submitted 2017-09-28; First posted 2018-12-19 (Actual); Last update posted 2018-12-27 (Actual); Status verified 2018-12

CONDITIONS: Resistance Training; Cardiovascular Risk; Low Birth Weight

STUDY DESIGN:
Intervention Model Description: The study is divided into two phases carried out in several visits: Phase I is constituted by a visit -1 and 1, which includes the selection of the sample and the randomization. Phase II includes the execution of the study with three arms, one group will be assigned to strength training and the other to aerobic capacity training, taking into account the plan of sessions per week defined for SIMAC (three sessions). The control group will be monitored passively for the detection of adverse or secondary events. At the end of this phase, anthropometric, clinical and biochemical markers will be monitored in the two intervention groups and in the control group. In Phase III a combined program of strength and aerobic capacity will be implemented, which will last six months more than will be compared with the previously defined control group.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The person responsible for the analyzes will be blind about the interventions. The analysis will be by intention to treat. There would be three arms of the study (strength group, aerobic exercise group and control group) of adolescents of 12 to 17 years old. A balanced randomization will be carried out using random numbers generated in software systematized form, guaranteeing the homogeneity of the number of subjects in each arm, with internal random assignment with a ratio of 1:1:1 to receive the study intervention.
Oversight: Data Monitoring Committee: No

ARMS (3):
- Habitual training (Active Comparator): The control group will be monitored passively for the detection of adverse or secondary events.
  Interventions: Behavioral: Muscular Resistance training; Behavioral: Cardiorespiratory training
- Muscular resistance training (Experimental): This phase includes the execution of the study with three arms, one group will be assigned to strength training and the other to aerobic capacity training, taking into account the plan of sessions per week.
  Interventions: Behavioral: Habitual training
- Cardiorespiratory training (Experimental): In stage, a combined program of strength and aerobic capacity will be implemented, which will last six months more than will be compared with the previously defined control group.
  Interventions: Behavioral: Habitual training

INTERVENTIONS:
Behavioral: Muscular Resistance training
  Arms: Habitual training
Behavioral: Cardiorespiratory training
  Arms: Habitual training
Behavioral: Habitual training
  Arms: Cardiorespiratory training; Muscular resistance training

SUMMARY:
Background Risk factors for cardiometabolic diseases have their onset in infancy. Comorbidities such as overweight, abdominal obesity, hypertension, insulin resistance and elevated triglycerides have been observed in childhood with a tendency to persist into adult life. Furthermore, this situation has generated an increase in morbidity and mortality rates due to chronic non-communicable diseases. One approach to decrease the impact of cardiometabolic diseases is the intervention with exercise training (strength and aerobic capacity), where an important role of protein intake plays a role in influencing the performance of strength training, due to the greater utilization of low-energy protein compared to aerobic exercise. In children, a better tolerance was reported in muscle strength exercises, with at least one supervised training session per week with moderate intensity (20 minutes of physical activity). Currently, there is no consensus on the minimum time required to intervene and achieve significant changes in the metabolic profile of adolescents and children.

Objective To evaluate the relationship between weight at birth and adaptations to aerobic exercise and muscular strength, and its effects on metabolic risk, body composition and physical capacity.

Methodology An experimental study with individual analysis per participant would be perform. The sample will include a 12 to 17-year-old adolescent population. It will consist of two phases. The intervention will be based on moderate strength, power and resistance training programs, and/or moderate aerobic capacity exercise in circuit steps. The workouts will be done two times a week, approximately 30 to 40 minutes including warm-up, stretching and cooling. All participants personal and family history data would be collected and blood samples would be taken.

Potential results Within the expected results, the protocol wants to implement a new methodology of physical capacity training. Furthermore, the protocol will evaluate if related cardiometabolic risk factors with the intervention would improve in target patients at risk of developing cardiometabolic diseases to identify them and prevent the occurrence of these pathologies in adult life.

DETAILED DESCRIPTION:
Type of study: Experimental study with individual analysis. Population object and sample: Adolescents from 12 to 17 years old of high school located in Bucaramanga's metropolitan area. The sample size was calculated to evaluate the difference between the maximum oxygen consumption (VO2max) between the control group and 20% of the intervention groups using an ANCOVA method, with a correlation of 0.5 between the initial and final evaluations. An error alpha of 0.05 and power of 0.8, obtaining a sample of 60 adolescents for each group.

Description of the physical intervention or program: This is a strength, power and endurance training program of moderate intensity combined with aerobic capacity training Moderate in the form of circuit. The trainings will be performed twice a week between 30-60 minutes of training, 1 hour including heating, stretching, explanations and cooling.

Baseline assessment: All adolescents will be provided with a CRF for past medical history and family history, a review of systems and physical examination. In addition, the following evaluation protocol is established: Health related physical fitness measurement (AFRS): Aerobic capacity, maximal strength, 6RM submaximal strength test, strength, power, muscular endurance and flexibility; Anthropometric measurements and body composition; Complete Blood Count (CBC), and Lipid Profile. Measurements with AFRS will be taken at baseline, after 3 months of the program and at the end (6 months).

Aerobic capacity: To measure the aerobic capacity, 20 Meter Shuttle Run Test will be applied. A site would be selected for the test, preferably a space of 25 meter or longer. It would need 4 cones, tape measure, compact disc (CD) with the test protocol and a CD player. The two ends of the 20-meter track should be clearly marked. For the execution, the adolescent will move from one line to another located 20 meters away and making the change of direction to the rhythm that is indicated by a sound signal that will progressively accelerate. The initial velocity of the signal would be 8.5 km/hr, and will increase by 0.5 km/hr/min (1 minute is equal to one shuttle). The test will end when the adolescent is not able to arrive for the second time in a row to the start line with the audio signal. Otherwise, the test will end when the teen stops because of fatigue. The participant would start running when the CD player emits the sound. The participant will touch the line at the end of the track with the feet, turn abruptly and run in the opposite direction. At first the speed will be low, but it will increase slowly and steadily every minute. The participant will stop when they no longer can keep the pace set. Or if they feel unable to complete the one-minute period. It is important to remember the last number announced by the CD player when the participant stops, because this will be the participant's score. This test would be performed only once. When the schoolchildren finish the test or cannot keep the pace, the last completed palier would be recorded.

Maximum isometric force: Hand dynamometry is an important test for assessing the physical performance and nutritional status of the participants and allows reference to the isometric muscular strength of the hand. The improve in muscle strengths are inversely associated with changes in total adiposity in childhood and adolescence. This test requires an adjustable dynamometer (TKK 5101 Grip D; Takey, Tokyo Japan) and a Right- and left-Hand Grip Rule. The Adolescent will tighten the dynamometer gradually and continuously for less than 2 seconds, performing the test twice (alternately with both hands) with the optimal grip adjustment according to the size of the hand (previously calculated with the hand grip rule). Allowing a short break between measurements for each measurement. The elbow should be in all its extension and the participant has to avoid the contact of the dynamometer with any part of the body. The Adolescent will take the dynamometer with one hand, try to apply the mayor strength possible. Would Squeeze gradually and continuously for less than 2 or 3 seconds. The examiner will show the correct form of execution. Adjust the grip measure according the size of the hand. The test will be done twice and the best result will be recorded. The maximum duration of the test will be 3-5 seconds, the size of the hand (right or left) should be measured to the maximum width. The accuracy of the measurement is 0.5 cm. During the test, the arm and hand holding the dynamometer do not touch the body. The instrument is held in line with the forearm. After a short break, a second attempt will be made.

Power: Vertical Jump Test is a test that measures the length reached in the vertical jump and with the Lewis's formula can calculate the power of the Adolescent. In addition, the participants can measure the force of the jump with a Platform Kinetics. To use it, the adolescent must stand at a side of a wall, and bring the hand closer to the wall, keeping their feet on the platform. They would have to jump vertically as high as possible with both legs. The platform kinetics would record the best of the three attempts. The participant must put the hands by the hips, to isolate the muscles of the legs. And three attempts are made to allow the coordination of arm movements. The vertical jump test is performed against a movement, where there is flexion of the knees before the jump. The necessary equipment to carry out this activity is the force plate (PASCO, USA, software, NMP technologies, London, UK).

Explosive force: The long jump test allows to measure muscle strength. For the test is needed a non-slip surface, a tape measure, tape and cones. The teenager is going to stand behind the jump line, they must stand with their feet in an equal distance to the anchor of their shoulders, parallel to the ground. Subsequently they will bend the knees with the arms in front of the body and from that position they will balance the arms, they will push with force and jump as far as possible. they will land on both feet simultaneously and in an upright position. The examiner will show the correct form of execution; the test will be done twice and the best result will be recorded. The horizontal lines of measurement are drawn in the drop landing zone at 10 cm, from 1 m from the take-off line. A tape measure is going to be put perpendicular to these lines. The examiner would be remained by the tape measure and will record the distance jumped by the adolescent. The jumped distance will be measured from the takeoff line to the back of the heel nearest to that line. A new attempt is allowed if the teenager falls backwards or contacts the surface with another part of the body.

Strength of resistance: Using the same test and the high jump protocol, but the participants would have to jump repeatedly for 15 seconds. The test is implemented with a Platform that allows the evaluation of the time in flight, time of contact between jumps and the power in each jump. The resistance is calculated with the average of these variables for 15 seconds and a fatigue index.

6-RM submaximal strength test: The American Academy of Pediatrics recommends strength training in the adolescent with a load adjusted to the ability of the Adolescent and with 6 maximal repetitions (6RM), which means that loading in an exercise should allow adolescents achieve 6 concentric and eccentric movements with good technique. In the program use a range of loads (RM's) It is going to be lighter adjusted to the assessment of the beginning of the program, and after every 6 weeks of training, the protocol will implement the test of 6 RM in exercise in machines (chest press, folding, shoulder press, extension of the Leg) to adjust the load according to the progression of the strength of each adolescent.

Flexibility: The protocol can define flexibility as the ability of the individual to get his/her body placed in as many positions as possible, both statics and moving positions. This implies a great capacity of mobility of the different corporal segments with an ample freedom of corporal movements.

Weight: The adolescent would be placed in the center of the scale in a standard upright position, without the body being in contact with anything around him/her. The participant will remain in the described position on the previously calibrated weight balance and it would be determined the weight in Kilograms.

Size: Have the participant stand erect on the floor board of the stadiometer with his or her back to the vertical backboard of the stadiometer. The weight of the participant is evenly distributed on both feet. The heels of the feet are placed together with both heels touching the base of the vertical board. Place the feet pointed slightly outward at a 60-degree angle. The adolescent will remain standing, keeping the position of Anthropometric attention with the heels, glutes, back and occipital region in contact with the vertical plane of the tallimeter. The evaluator makes an in-depth inspiration at the time of the measurement to compensate for the shortening of the intervertebral discs.

Body mass index - BMI: The body mass index or the Quetelet index, has been defined as the ratio of weight to height squared (kilogram/m2). This index changes substantially with age, at birth, is as low as 13 kg/m2. The CDC proposes to use as cutoffs of the 85th and 95th percentile of its own data.

Development of the study: There would be three arms of the study (strength group, aerobic exercise group and control group) of adolescents of 12 to 17 years old. The person responsible for the analyzes will be blind about the interventions. The analysis will be by intention to treat. Once the inclusion/exclusion criteria are checked, the selected candidates will receive information about the study objectives and methodology, and finally the adolescent will sign the informed consent and the guardian or responsible of the child will sign the informed consent too. After the screening procedures and the initial evaluation of the inclusion and selection criteria, the patients will begin the initial evaluation period. A balanced randomization will be carried out using random numbers generated in software systematized form, guaranteeing the homogeneity of the number of subjects in each arm, with internal random assignment with a ratio of 1:1:1 to receive the study intervention. This study is designed with a primary efficacy endpoint at six months and at twelve months. Upon completion of 6 months of intervention, the strength and aerobic capacity groups would be integrated into a single group to evaluate the combined effect of the interventions versus the control group.

The study is divided into two phases carried out in several visits: Phase I is constituted by a visit -1 and 1, which includes the selection of the sample and the randomization. Phase II includes the execution of the study with three arms, one group will be assigned to strength training and the other to aerobic capacity training, taking into account the plan of sessions per week defined for SIMAC (three sessions). The control group will be monitored passively for the detection of adverse or secondary events. At the end of this phase, anthropometric, clinical and biochemical markers will be monitored in the two intervention groups and in the control group. In Phase III a combined program of strength and aerobic capacity will be implemented, which will last six months more than will be compared with the previously defined control group. Again, at the end of phase III, the outcomes related to possible changes in the anthropometric, clinical and biochemical markers in the two groups will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents 12-17 years old.
* Tanner 3 at medical evaluation.
* Provide reliable information on birth weight and gestational age.
* For the group of Low birth weight: birth weight below 2800 gr. For the group of normal birth weight: birth weight between 2800 - 4000 gr

Exclusion Criteria:

* Express voluntarily desire for non-participation by parents in the study.
* Teenager's desire of not to be included in the study.
* Adolescents with physical disability that prevents them from engaging in a physical training program focused on strengthening.
* Adolescents with asthma.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 150 (Actual)
Dates: Start 2016-02-01; Primary Completion 2016-07-30 (Actual); Study Completion 2016-12-10 (Actual)

PRIMARY OUTCOMES:
% of change in the glucose levels within the experimental groups with the habitual training | Twelve months
  Evaluation of cardiometabolic risk factors related to physical training to take into account in patients with a risk of developing cardiometabolic diseases and that have as antecedents low birth weight to identify them and prevent the appearance of these pathologies that affect the health and quality of life
% of change in the body mass index within the experimental groups with the habitual training | Twelve months
  Evaluation of cardiometabolic risk factors related to physical training to take into account in patients with a risk of developing cardiometabolic diseases and that have as antecedents low birth weight to identify them and prevent the appearance of these pathologies that affect the health and quality of life
% of change in the lipid profile levels within the experimental groups with the habitual training | Twelve months
  Evaluation of cardiometabolic risk factors related to physical training to take into account in patients with a risk of developing cardiometabolic diseases and that have as antecedents low birth weight to identify them and prevent the appearance of these pathologies that affect the health and quality of life

SECONDARY OUTCOMES:
% change in the hand grip strenght test within the experimental groups with the habitual training | Twelve months
  % change in physical fitness in the participants of the experimental group compared to the control group in hand grip strenght test , as markers of cardiometabolic risk (glucose, lipid profile and body mass index)
% change in the flexibility within the experimental groups with the habitual training | Twelve months
  % change in physical fitness in the participants of the experimental group compared to the control group in flexibility with sit and reach, as markers of cardiometabolic risk (glucose, lipid profile and BMI)
% change in the vertical jump within the experimental groups with the habitual training | Twelve months
  % change in physical fitness in the participants of the experimental group compared to the control group in vertical jump, as markers of cardiometabolic risk (glucose, lipid profile and BMI)

CONTACTS AND LOCATIONS:
Overall Officials: PATRICIO LOPEZ, JARAMILLO, Study Director — FUNDACION OFTALMOLOGICA DE SANTANDER

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cohen DD, Gomez-Arbelaez D, Camacho PA, Pinzon S, Hormiga C, Trejos-Suarez J, Duperly J, Lopez-Jaramillo P. Low muscle strength is associated with metabolic risk factors in Colombian children: the ACFIES study. PLoS One. 2014 Apr 8;9(4):e93150. doi: 10.1371/journal.pone.0093150. eCollection 2014. PMID 24714401
- [Background] Raitakari OT, Juonala M, Kahonen M, Taittonen L, Laitinen T, Maki-Torkko N, Jarvisalo MJ, Uhari M, Jokinen E, Ronnemaa T, Akerblom HK, Viikari JS. Cardiovascular risk factors in childhood and carotid artery intima-media thickness in adulthood: the Cardiovascular Risk in Young Finns Study. JAMA. 2003 Nov 5;290(17):2277-83. doi: 10.1001/jama.290.17.2277. PMID 14600186
- [Background] Lopez-Jaramillo P. Cardiometabolic disease in latin america: the role of fetal programming in response to maternal malnutrition. Rev Esp Cardiol. 2009 Jun;62(6):670-6. doi: 10.1016/s1885-5857(09)72231-5. English, Spanish. PMID 19480763
- [Background] Steene-Johannessen J, Anderssen SA, Kolle E, Andersen LB. Low muscle fitness is associated with metabolic risk in youth. Med Sci Sports Exerc. 2009 Jul;41(7):1361-7. doi: 10.1249/MSS.0b013e31819aaae5. PMID 19516166
- [Background] Lopez-Jaramillo P. Defining the research priorities to fight the burden of cardiovascular diseases in Latin America. J Hypertens. 2008 Sep;26(9):1886-9. doi: 10.1097/HJH.0b013e328308ba8d. No abstract available. PMID 18698226
- [Background] OMS OMdlS-. Estrategia mundial sobre régimen alimentario, actividad física y salud. [updated 12-06-2014; cited 2014 12-06-2014]; Available from: http://www.who.int/dietphysicalactivity/childhood/es/.
- [Background] Benson AC, Torode ME, Singh MA. Muscular strength and cardiorespiratory fitness is associated with higher insulin sensitivity in children and adolescents. Int J Pediatr Obes. 2006;1(4):222-31. doi: 10.1080/17477160600962864. PMID 17907329
- [Background] Lopez-Jaramillo P, Lahera V, Lopez-Lopez J. Epidemic of cardiometabolic diseases: a Latin American point of view. Ther Adv Cardiovasc Dis. 2011 Apr;5(2):119-31. doi: 10.1177/1753944711403189. Epub 2011 Mar 15. PMID 21406494
- [Background] Lopez-Jaramillo P, Silva SY, Rodriguez-Salamanca N, Duran A, Mosquera W, Castillo V. Are nutrition-induced epigenetic changes the link between socioeconomic pathology and cardiovascular diseases? Am J Ther. 2008 Jul-Aug;15(4):362-72. doi: 10.1097/MJT.0b013e318164bf9c. PMID 18645341
- [Background] López-Jaramillo P, López-López J. Fetal programming and cardiometabolic diseases: the role of angiotensin II and inflammation. Clínica e Investigación en Arteriosclerosis. 2010;22, Supplement 2(0):21-4.
- [Background] Yusuf S, Hawken S, Ounpuu S, Dans T, Avezum A, Lanas F, McQueen M, Budaj A, Pais P, Varigos J, Lisheng L; INTERHEART Study Investigators. Effect of potentially modifiable risk factors associated with myocardial infarction in 52 countries (the INTERHEART study): case-control study. Lancet. 2004 Sep 11-17;364(9438):937-52. doi: 10.1016/S0140-6736(04)17018-9. PMID 15364185
- [Background] Lanas F, Avezum A, Bautista LE, Diaz R, Luna M, Islam S, Yusuf S; INTERHEART Investigators in Latin America. Risk factors for acute myocardial infarction in Latin America: the INTERHEART Latin American study. Circulation. 2007 Mar 6;115(9):1067-74. doi: 10.1161/CIRCULATIONAHA.106.633552. PMID 17339564
- [Background] Gomez-Arbelaez D, Camacho PA, Cohen DD, Rincon-Romero K, Alvarado-Jurado L, Pinzon S, Duperly J, Lopez-Jaramillo P. Higher household income and the availability of electronic devices and transport at home are associated with higher waist circumference in Colombian children: the ACFIES study. Int J Environ Res Public Health. 2014 Feb 7;11(2):1834-43. doi: 10.3390/ijerph110201834. PMID 24514426
- [Background] López Jaramillo P, Gómez Arbeláez D, Cohen DD, Camacho PA, Rincón Romero K, Hormiga C, et al. Association between obesity and low muscular and cardiorespiratory capacity, cardiometabolic risk factors in Colombian children. Trauma. 2013;24(1):17-23.
- [Background] Lopez-Jaramillo P, Herrera E, Garcia RG, Camacho PA, Castillo VR. Inter-relationships between body mass index, C-reactive protein and blood pressure in a Hispanic pediatric population. Am J Hypertens. 2008 May;21(5):527-32. doi: 10.1038/ajh.2007.86. Epub 2008 Mar 6. PMID 18437144
- [Background] Tresierras MA, Balady GJ. Resistance training in the treatment of diabetes and obesity: mechanisms and outcomes. J Cardiopulm Rehabil Prev. 2009 Mar-Apr;29(2):67-75. doi: 10.1097/HCR.0b013e318199ff69. PMID 19305230
- [Background] Faigenbaum AD, Westcott WL, Loud RL, Long C. The effects of different resistance training protocols on muscular strength and endurance development in children. Pediatrics. 1999 Jul;104(1):e5. doi: 10.1542/peds.104.1.e5. PMID 10390291
- [Background] Faigenbaum AD, Milliken LA, Loud RL, Burak BT, Doherty CL, Westcott WL. Comparison of 1 and 2 days per week of strength training in children. Res Q Exerc Sport. 2002 Dec;73(4):416-24. doi: 10.1080/02701367.2002.10609041. PMID 12495243
- [Background] Malina RM. Weight training in youth-growth, maturation, and safety: an evidence-based review. Clin J Sport Med. 2006 Nov;16(6):478-87. doi: 10.1097/01.jsm.0000248843.31874.be. PMID 17119361
- [Background] Pikosky M, Faigenbaum A, Westcott W, Rodriguez N. Effects of resistance training on protein utilization in healthy children. Med Sci Sports Exerc. 2002 May;34(5):820-7. doi: 10.1097/00005768-200205000-00015. PMID 11984301
- [Background] Shaibi GQ, Cruz ML, Ball GD, Weigensberg MJ, Salem GJ, Crespo NC, Goran MI. Effects of resistance training on insulin sensitivity in overweight Latino adolescent males. Med Sci Sports Exerc. 2006 Jul;38(7):1208-15. doi: 10.1249/01.mss.0000227304.88406.0f. PMID 16826016
- [Background] Holten MK, Zacho M, Gaster M, Juel C, Wojtaszewski JF, Dela F. Strength training increases insulin-mediated glucose uptake, GLUT4 content, and insulin signaling in skeletal muscle in patients with type 2 diabetes. Diabetes. 2004 Feb;53(2):294-305. doi: 10.2337/diabetes.53.2.294. PMID 14747278
- [Background] Bell LM, Watts K, Siafarikas A, Thompson A, Ratnam N, Bulsara M, Finn J, O'Driscoll G, Green DJ, Jones TW, Davis EA. Exercise alone reduces insulin resistance in obese children independently of changes in body composition. J Clin Endocrinol Metab. 2007 Nov;92(11):4230-5. doi: 10.1210/jc.2007-0779. Epub 2007 Aug 14. PMID 17698905
- [Background] Moore DR, Del Bel NC, Nizi KI, Hartman JW, Tang JE, Armstrong D, Phillips SM. Resistance training reduces fasted- and fed-state leucine turnover and increases dietary nitrogen retention in previously untrained young men. J Nutr. 2007 Apr;137(4):985-91. doi: 10.1093/jn/137.4.985. PMID 17374665
- [Background] Mascher H, Tannerstedt J, Brink-Elfegoun T, Ekblom B, Gustafsson T, Blomstrand E. Repeated resistance exercise training induces different changes in mRNA expression of MAFbx and MuRF-1 in human skeletal muscle. Am J Physiol Endocrinol Metab. 2008 Jan;294(1):E43-51. doi: 10.1152/ajpendo.00504.2007. Epub 2007 Oct 30. PMID 17971512
- [Background] Ballor DL, Katch VL, Becque MD, Marks CR. Resistance weight training during caloric restriction enhances lean body weight maintenance. Am J Clin Nutr. 1988 Jan;47(1):19-25. doi: 10.1093/ajcn/47.1.19. PMID 3337037
- [Background] Kraemer WJ, Volek JS, Clark KL, Gordon SE, Puhl SM, Koziris LP, McBride JM, Triplett-McBride NT, Putukian M, Newton RU, Hakkinen K, Bush JA, Sebastianelli WJ. Influence of exercise training on physiological and performance changes with weight loss in men. Med Sci Sports Exerc. 1999 Sep;31(9):1320-9. doi: 10.1097/00005768-199909000-00014. PMID 10487375
- [Background] Faigenbaum AD, Kraemer WJ, Blimkie CJ, Jeffreys I, Micheli LJ, Nitka M, Rowland TW. Youth resistance training: updated position statement paper from the national strength and conditioning association. J Strength Cond Res. 2009 Aug;23(5 Suppl):S60-79. doi: 10.1519/JSC.0b013e31819df407. PMID 19620931
- [Background] American Academy of Pediatrics Council on Sports Medicine and Fitness; McCambridge TM, Stricker PR. Strength training by children and adolescents. Pediatrics. 2008 Apr;121(4):835-40. doi: 10.1542/peds.2007-3790. PMID 18381549
- [Background] Popkin BM. The nutrition transition: an overview of world patterns of change. Nutr Rev. 2004 Jul;62(7 Pt 2):S140-3. doi: 10.1111/j.1753-4887.2004.tb00084.x. PMID 15387480
- [Background] Lopez P. Capítulo 1: Las enfermedades Cardiovasculares en los países subdesarrollados Bioquímica del endotelio vascular: Implicaciones fisiológicas y clínicas 2001. p. 21 - 34.
- [Background] Barker DJ, Meade TW, Fall CH, Lee A, Osmond C, Phipps K, Stirling Y. Relation of fetal and infant growth to plasma fibrinogen and factor VII concentrations in adult life. BMJ. 1992 Jan 18;304(6820):148-52. doi: 10.1136/bmj.304.6820.148. PMID 1737158
- [Background] Victora CG, Adair L, Fall C, Hallal PC, Martorell R, Richter L, Sachdev HS; Maternal and Child Undernutrition Study Group. Maternal and child undernutrition: consequences for adult health and human capital. Lancet. 2008 Jan 26;371(9609):340-57. doi: 10.1016/S0140-6736(07)61692-4. PMID 18206223
- [Background] Prentice AM, Moore SE. Early programming of adult diseases in resource poor countries. Arch Dis Child. 2005 Apr;90(4):429-32. doi: 10.1136/adc.2004.059030. PMID 15781942
- [Background] Wright CM, Parker L, Lamont D, Craft AW. Implications of childhood obesity for adult health: findings from thousand families cohort study. BMJ. 2001 Dec 1;323(7324):1280-4. doi: 10.1136/bmj.323.7324.1280. PMID 11731390
- [Background] Sawaya AL, Dallal G, Solymos G, de Sousa MH, Ventura ML, Roberts SB, Sigulem DM. Obesity and malnutrition in a Shantytown population in the city of Sao Paulo, Brazil. Obes Res. 1995 Sep;3 Suppl 2:107s-115s. doi: 10.1002/j.1550-8528.1995.tb00453.x. PMID 8581766
- [Background] Black RE, Victora CG, Walker SP, Bhutta ZA, Christian P, de Onis M, Ezzati M, Grantham-McGregor S, Katz J, Martorell R, Uauy R; Maternal and Child Nutrition Study Group. Maternal and child undernutrition and overweight in low-income and middle-income countries. Lancet. 2013 Aug 3;382(9890):427-451. doi: 10.1016/S0140-6736(13)60937-X. Epub 2013 Jun 6. PMID 23746772
- [Background] Perez-Farinos N, Lopez-Sobaler AM, Dal Re MA, Villar C, Labrado E, Robledo T, Ortega RM. The ALADINO study: a national study of prevalence of overweight and obesity in Spanish children in 2011. Biomed Res Int. 2013;2013:163687. doi: 10.1155/2013/163687. Epub 2013 Sep 8. PMID 24089663
- [Background] Touwslager RN, Gielen M, Tan FE, Mulder AL, Gerver WJ, Zimmermann LJ, Houben AJ, Zeegers MP, Derom C, Vlietinck R, Maes HH, Stehouwer CD, Thomis M. Genetic, maternal and placental factors in the association between birth weight and physical fitness: a longitudinal twin study. PLoS One. 2013 Oct 23;8(10):e76423. doi: 10.1371/journal.pone.0076423. eCollection 2013. PMID 24194838
- [Background] Kuh D, Bassey J, Hardy R, Aihie Sayer A, Wadsworth M, Cooper C. Birth weight, childhood size, and muscle strength in adult life: evidence from a birth cohort study. Am J Epidemiol. 2002 Oct 1;156(7):627-33. doi: 10.1093/aje/kwf099. PMID 12244031
- [Background] Inskip HM, Godfrey KM, Martin HJ, Simmonds SJ, Cooper C, Sayer AA; Southampton Women's Survey Study Group. Size at birth and its relation to muscle strength in young adult women. J Intern Med. 2007 Sep;262(3):368-74. doi: 10.1111/j.1365-2796.2007.01812.x. PMID 17697158
- [Background] Ortega FB, Ruiz JR, Labayen I, Redondo C, Breidenassel C, Gomez S, Moreno LA, Castillo MJ; Avena Study Group. High fitness is associated with a healthier programming of body composition at adolescence. Am J Hum Biol. 2008 Nov-Dec;20(6):732-4. doi: 10.1002/ajhb.20813. PMID 18770529
- [Background] Laaksonen DE, Lakka HM, Lynch J, Lakka TA, Niskanen L, Rauramaa R, Salonen JT, Kauhanen J. Cardiorespiratory fitness and vigorous leisure-time physical activity modify the association of small size at birth with the metabolic syndrome. Diabetes Care. 2003 Jul;26(7):2156-64. doi: 10.2337/diacare.26.7.2156. PMID 12832329
- [Background] Ortega FB, Artero EG, Ruiz JR, Espana-Romero V, Jimenez-Pavon D, Vicente-Rodriguez G, Moreno LA, Manios Y, Beghin L, Ottevaere C, Ciarapica D, Sarri K, Dietrich S, Blair SN, Kersting M, Molnar D, Gonzalez-Gross M, Gutierrez A, Sjostrom M, Castillo MJ; HELENA study. Physical fitness levels among European adolescents: the HELENA study. Br J Sports Med. 2011 Jan;45(1):20-9. doi: 10.1136/bjsm.2009.062679. Epub 2009 Aug 20. PMID 19700434
- [Background] Wells JC, Chomtho S, Fewtrell MS. Programming of body composition by early growth and nutrition. Proc Nutr Soc. 2007 Aug;66(3):423-34. doi: 10.1017/S0029665107005691. PMID 17637095
- [Background] Eriksson M, Tynelius P, Rasmussen F. Associations of birthweight and infant growth with body composition at age 15--the COMPASS study. Paediatr Perinat Epidemiol. 2008 Jul;22(4):379-88. doi: 10.1111/j.1365-3016.2008.00944.x. PMID 18578752
- [Background] Wells JC, Hallal PC, Wright A, Singhal A, Victora CG. Fetal, infant and childhood growth: relationships with body composition in Brazilian boys aged 9 years. Int J Obes (Lond). 2005 Oct;29(10):1192-8. doi: 10.1038/sj.ijo.0803054. PMID 16103893
- [Background] Kelly LA, Lane CJ, Ball GD, Weigensberg MJ, Vargas LG, Byrd-Williams CE, Ventura EE, Goran MI. Birth weight and body composition in overweight Latino youth: a longitudinal analysis. Obesity (Silver Spring). 2008 Nov;16(11):2524-8. doi: 10.1038/oby.2008.401. Epub 2008 Sep 11. PMID 18787529
- [Background] Sawaya AL, Martins P, Hoffman D, Roberts SB. The link between childhood undernutrition and risk of chronic diseases in adulthood: a case study of Brazil. Nutr Rev. 2003 May;61(5 Pt 1):168-75. doi: 10.1301/nr.2003.may.168-175. PMID 12822705
- [Background] Yajnik CS, Fall CH, Coyaji KJ, Hirve SS, Rao S, Barker DJ, Joglekar C, Kellingray S. Neonatal anthropometry: the thin-fat Indian baby. The Pune Maternal Nutrition Study. Int J Obes Relat Metab Disord. 2003 Feb;27(2):173-80. doi: 10.1038/sj.ijo.802219. PMID 12586996
- [Background] Sayer AA, Syddall HE, Gilbody HJ, Dennison EM, Cooper C. Does sarcopenia originate in early life? Findings from the Hertfordshire cohort study. J Gerontol A Biol Sci Med Sci. 2004 Sep;59(9):M930-4. doi: 10.1093/gerona/59.9.m930. PMID 15472158
- [Background] Jackson AW, Lee DC, Sui X, Morrow JR Jr, Church TS, Maslow AL, Blair SN. Muscular strength is inversely related to prevalence and incidence of obesity in adult men. Obesity (Silver Spring). 2010 Oct;18(10):1988-95. doi: 10.1038/oby.2009.422. Epub 2009 Dec 3. PMID 19960002
- [Background] Lazarus R, Sparrow D, Weiss ST. Handgrip strength and insulin levels: cross-sectional and prospective associations in the Normative Aging Study. Metabolism. 1997 Nov;46(11):1266-9. doi: 10.1016/s0026-0495(97)90228-6. PMID 9361683
- [Background] Silventoinen K, Magnusson PK, Tynelius P, Batty GD, Rasmussen F. Association of body size and muscle strength with incidence of coronary heart disease and cerebrovascular diseases: a population-based cohort study of one million Swedish men. Int J Epidemiol. 2009 Feb;38(1):110-8. doi: 10.1093/ije/dyn231. Epub 2008 Nov 25. PMID 19033357
- [Background] Ruiz JR, Sui X, Lobelo F, Lee DC, Morrow JR Jr, Jackson AW, Hebert JR, Matthews CE, Sjostrom M, Blair SN. Muscular strength and adiposity as predictors of adulthood cancer mortality in men. Cancer Epidemiol Biomarkers Prev. 2009 May;18(5):1468-76. doi: 10.1158/1055-9965.EPI-08-1075. Epub 2009 Apr 14. PMID 19366909
- [Background] Cruz-Jentoft AJ, Baeyens JP, Bauer JM, Boirie Y, Cederholm T, Landi F, Martin FC, Michel JP, Rolland Y, Schneider SM, Topinkova E, Vandewoude M, Zamboni M; European Working Group on Sarcopenia in Older People. Sarcopenia: European consensus on definition and diagnosis: Report of the European Working Group on Sarcopenia in Older People. Age Ageing. 2010 Jul;39(4):412-23. doi: 10.1093/ageing/afq034. Epub 2010 Apr 13. PMID 20392703
- [Background] Jensen CB, Martin-Gronert MS, Storgaard H, Madsbad S, Vaag A, Ozanne SE. Altered PI3-kinase/Akt signalling in skeletal muscle of young men with low birth weight. PLoS One. 2008;3(11):e3738. doi: 10.1371/journal.pone.0003738. Epub 2008 Nov 17. PMID 19011679
- [Background] Jensen CB, Storgaard H, Madsbad S, Richter EA, Vaag AA. Altered skeletal muscle fiber composition and size precede whole-body insulin resistance in young men with low birth weight. J Clin Endocrinol Metab. 2007 Apr;92(4):1530-4. doi: 10.1210/jc.2006-2360. Epub 2007 Feb 6. PMID 17284623
- [Background] Ozanne SE, Jensen CB, Tingey KJ, Storgaard H, Madsbad S, Vaag AA. Low birthweight is associated with specific changes in muscle insulin-signalling protein expression. Diabetologia. 2005 Mar;48(3):547-52. doi: 10.1007/s00125-005-1669-7. Epub 2005 Feb 24. PMID 15729577
- [Background] Scribbans TD, Edgett BA, Vorobej K, Mitchell AS, Joanisse SD, Matusiak JB, Parise G, Quadrilatero J, Gurd BJ. Fibre-specific responses to endurance and low volume high intensity interval training: striking similarities in acute and chronic adaptation. PLoS One. 2014 Jun 5;9(6):e98119. doi: 10.1371/journal.pone.0098119. eCollection 2014. PMID 24901767
- [Background] Bruce CR, Anderson MJ, Carey AL, Newman DG, Bonen A, Kriketos AD, Cooney GJ, Hawley JA. Muscle oxidative capacity is a better predictor of insulin sensitivity than lipid status. J Clin Endocrinol Metab. 2003 Nov;88(11):5444-51. doi: 10.1210/jc.2003-030791. PMID 14602787
- [Background] Olsson AH, Ronn T, Elgzyri T, Hansson O, Eriksson KF, Groop L, Vaag A, Poulsen P, Ling C. The expression of myosin heavy chain (MHC) genes in human skeletal muscle is related to metabolic characteristics involved in the pathogenesis of type 2 diabetes. Mol Genet Metab. 2011 Jul;103(3):275-81. doi: 10.1016/j.ymgme.2011.03.017. Epub 2011 Mar 21. PMID 21470888
- [Background] Wade AJ, Marbut MM, Round JM. Muscle fibre type and aetiology of obesity. Lancet. 1990 Apr 7;335(8693):805-8. doi: 10.1016/0140-6736(90)90933-v. PMID 1969558
- [Background] Tikkanen HO, Hamalainen E, Sarna S, Adlercreutz H, Harkonen M. Associations between skeletal muscle properties, physical fitness, physical activity and coronary heart disease risk factors in men. Atherosclerosis. 1998 Apr;137(2):377-89. doi: 10.1016/s0021-9150(97)00276-1. PMID 9622281
- [Background] Frosig C, Richter EA. Improved insulin sensitivity after exercise: focus on insulin signaling. Obesity (Silver Spring). 2009 Dec;17 Suppl 3:S15-20. doi: 10.1038/oby.2009.383. PMID 19927140
- [Background] Daugaard JR, Nielsen JN, Kristiansen S, Andersen JL, Hargreaves M, Richter EA. Fiber type-specific expression of GLUT4 in human skeletal muscle: influence of exercise training. Diabetes. 2000 Jul;49(7):1092-5. doi: 10.2337/diabetes.49.7.1092. PMID 10909963
- [Background] Simoneau JA, Lortie G, Boulay MR, Marcotte M, Thibault MC, Bouchard C. Human skeletal muscle fiber type alteration with high-intensity intermittent training. Eur J Appl Physiol Occup Physiol. 1985;54(3):250-3. doi: 10.1007/BF00426141. PMID 4065109
- [Background] Fry AC. The role of resistance exercise intensity on muscle fibre adaptations. Sports Med. 2004;34(10):663-79. doi: 10.2165/00007256-200434100-00004. PMID 15335243
- [Background] Miller BF, Olesen JL, Hansen M, Dossing S, Crameri RM, Welling RJ, Langberg H, Flyvbjerg A, Kjaer M, Babraj JA, Smith K, Rennie MJ. Coordinated collagen and muscle protein synthesis in human patella tendon and quadriceps muscle after exercise. J Physiol. 2005 Sep 15;567(Pt 3):1021-33. doi: 10.1113/jphysiol.2005.093690. Epub 2005 Jul 7. PMID 16002437
- [Background] Phillips SM, Tipton KD, Aarsland A, Wolf SE, Wolfe RR. Mixed muscle protein synthesis and breakdown after resistance exercise in humans. Am J Physiol. 1997 Jul;273(1 Pt 1):E99-107. doi: 10.1152/ajpendo.1997.273.1.E99. PMID 9252485
- [Background] Petersen AM, Pedersen BK. The anti-inflammatory effect of exercise. J Appl Physiol (1985). 2005 Apr;98(4):1154-62. doi: 10.1152/japplphysiol.00164.2004. PMID 15772055
- [Background] Shaibi GQ, Cruz ML, Weigensberg MJ, Toledo-Corral CM, Lane CJ, Kelly LA, Davis JN, Koebnick C, Ventura EE, Roberts CK, Goran MI. Adiponectin independently predicts metabolic syndrome in overweight Latino youth. J Clin Endocrinol Metab. 2007 May;92(5):1809-13. doi: 10.1210/jc.2006-2294. Epub 2007 Feb 20. PMID 17311859
- [Background] Nappo A, Iacoviello L, Fraterman A, Gonzalez-Gil EM, Hadjigeorgiou C, Marild S, Molnar D, Moreno LA, Peplies J, Sioen I, Veidebaum T, Siani A, Russo P. High-sensitivity C-reactive protein is a predictive factor of adiposity in children: results of the identification and prevention of dietary- and lifestyle-induced health effects in children and infants (IDEFICS) study. J Am Heart Assoc. 2013 Jun 6;2(3):e000101. doi: 10.1161/JAHA.113.000101. PMID 23744403
- [Background] Nazmi A, Victora CG. Socioeconomic and racial/ethnic differentials of C-reactive protein levels: a systematic review of population-based studies. BMC Public Health. 2007 Aug 17;7:212. doi: 10.1186/1471-2458-7-212. PMID 17705867
- [Background] Ruiz JR, Ortega FB, Warnberg J, Moreno LA, Carrero JJ, Gonzalez-Gross M, Marcos A, Gutierrez A, Sjostrom M. Inflammatory proteins and muscle strength in adolescents: the Avena study. Arch Pediatr Adolesc Med. 2008 May;162(5):462-8. doi: 10.1001/archpedi.162.5.462. PMID 18458193
- [Background] Donges CE, Duffield R, Drinkwater EJ. Effects of resistance or aerobic exercise training on interleukin-6, C-reactive protein, and body composition. Med Sci Sports Exerc. 2010 Feb;42(2):304-13. doi: 10.1249/MSS.0b013e3181b117ca. PMID 20083961
- [Background] Daray LA, Henagan TM, Zanovec M, Earnest CP, Johnson LG, Winchester J, Tuuri G, Stewart LK. Endurance and resistance training lowers C-reactive protein in young, healthy females. Appl Physiol Nutr Metab. 2011 Oct;36(5):660-70. doi: 10.1139/h11-077. Epub 2011 Oct 4. PMID 21970447
- [Background] Kamal NN, Ragy MM. The effects of exercise on C-reactive protein, insulin, leptin and some cardiometabolic risk factors in Egyptian children with or without metabolic syndrome. Diabetol Metab Syndr. 2012 Jun 12;4(1):27. doi: 10.1186/1758-5996-4-27. PMID 22691465
- [Background] Nassis GP, Papantakou K, Skenderi K, Triandafillopoulou M, Kavouras SA, Yannakoulia M, Chrousos GP, Sidossis LS. Aerobic exercise training improves insulin sensitivity without changes in body weight, body fat, adiponectin, and inflammatory markers in overweight and obese girls. Metabolism. 2005 Nov;54(11):1472-9. doi: 10.1016/j.metabol.2005.05.013. PMID 16253636
- [Background] Artero EG, Lee DC, Lavie CJ, Espana-Romero V, Sui X, Church TS, Blair SN. Effects of muscular strength on cardiovascular risk factors and prognosis. J Cardiopulm Rehabil Prev. 2012 Nov-Dec;32(6):351-8. doi: 10.1097/HCR.0b013e3182642688. PMID 22885613
- [Background] Lopez-Jaramillo P, Cohen DD, Gomez-Arbelaez D, Bosch J, Dyal L, Yusuf S, Gerstein HC; ORIGIN Trial Investigators. Association of handgrip strength to cardiovascular mortality in pre-diabetic and diabetic patients: a subanalysis of the ORIGIN trial. Int J Cardiol. 2014 Jun 15;174(2):458-61. doi: 10.1016/j.ijcard.2014.04.013. Epub 2014 Apr 13. No abstract available. PMID 24768457
- [Background] van Deutekom AW, Chinapaw MJ, Vrijkotte TG, Gemke RJ. Study protocol: the relation of birth weight and infant growth trajectories with physical fitness, physical activity and sedentary behavior at 8-9 years of age - the ABCD study. BMC Pediatr. 2013 Jul 9;13:102. doi: 10.1186/1471-2431-13-102. PMID 23835159
- [Background] Ridgway CL, Brage S, Anderssen S, Sardinha LB, Andersen LB, Ekelund U. Fat-free mass mediates the association between birth weight and aerobic fitness in youth. Int J Pediatr Obes. 2011 Jun;6(2-2):e590-6. doi: 10.3109/17477166.2010.526225. Epub 2010 Nov 4. PMID 21050079
- [Background] Brons C, Jensen CB, Storgaard H, Alibegovic A, Jacobsen S, Nilsson E, Astrup A, Quistorff B, Vaag A. Mitochondrial function in skeletal muscle is normal and unrelated to insulin action in young men born with low birth weight. J Clin Endocrinol Metab. 2008 Oct;93(10):3885-92. doi: 10.1210/jc.2008-0630. Epub 2008 Jul 15. PMID 18628517
- [Background] Batería ALPHA-Fitness: Test de campo para la evaluación de la condición física relacionada con la salud en niños y adolescentes.Pag 21
- [Background] Tremblay MS, Shields M, Laviolette M, Craig CL, Janssen I, Connor Gorber S. Fitness of Canadian children and youth: results from the 2007-2009 Canadian Health Measures Survey. Health Rep. 2010 Mar;21(1):7-20. PMID 20426223
- [Background] Cohen DD, Voss C, Taylor MJ, Stasinopoulos DM, Delextrat A, Sandercock GR. Handgrip strength in English schoolchildren. Acta Paediatr. 2010 Jul;99(7):1065-72. doi: 10.1111/j.1651-2227.2010.01723.x. Epub 2010 Feb 19. PMID 20178516
- [Background] Marrodan Serrano MD, Romero Collazos JF, Moreno Romero S, Mesa Santurino MS, Cabanas Armesilla MD, Pacheco Del Cerro JL, Gonzalez-Montero de Espinosa M. [Handgrip strength in children and teenagers aged from 6 to 18 years: reference values and relationship with size and body composition]. An Pediatr (Barc). 2009 Apr;70(4):340-8. doi: 10.1016/j.anpedi.2008.11.025. Epub 2009 Mar 5. Spanish. PMID 19268640
- [Background] RICKE O, SCHOENAU E ibid Pag 228
- [Background] ESCALONA P, NARANJO J,LAGOS V, SOLÍS F. Normal Parameters in Hand Grasping Strength in subjects of both genders, 7 to 17 years of age. Rev Chil Pediatr 2009; 80 (5): 435-443
- [Background] FLORES-HUERTA S. Antropometría, estado nutricio y salud de los niños. Importancia de las mediciones comparables. Bol Med Hosp Infant Mex. Vol. 63, Marzo-Abril 2006. Pag. 74.
- [Background] Fuller NJ, Fewtrell MS, Dewit O, Elia M, Wells JC. Segmental bioelectrical impedance analysis in children aged 8-12 y: 2. The assessment of regional body composition and muscle mass. Int J Obes Relat Metab Disord. 2002 May;26(5):692-700. doi: 10.1038/sj.ijo.0801989. PMID 12032755
- [Background] Kilani H, Abu-Eisheh A. Optimum anthropometric criteria for ideal body composition related fitness. Sultan Qaboos Univ Med J. 2010 Apr;10(1):74-9. Epub 2010 Apr 17. PMID 21509084